CLINICAL TRIAL: NCT03241173
Title: A Phase 1/2 Study Exploring the Safety, Tolerability, and Efficacy of INCAGN01949 in Combination With Immune Therapies in Subjects With Advanced or Metastatic Malignancies
Brief Title: A Study Exploring the Safety and Efficacy of INCAGN01949 in Combination With Immune Therapies in Advanced or Metastatic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 1949-201
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Advanced Malignancies
Keywords: advanced or metastatic cervical cancer; endometrial cancer; esophageal cancer; hepatocellular carcinoma (HCC); melanoma; Merkel cell carcinoma; mesothelioma; microsatellite instability-high colorectal cancer; non-small cell lung cancer (NSCLC); ovarian cancer; squamous cell carcinoma of the head and neck; small cell lung cancer (SLCL); renal cell carcinoma (RCC); triple-negative breast cancer; TNBC; urothelial carcinoma; OX40 ligand (OX40); SCCHN; MSI-H CRC; gastric cancer (including stomach and gastroesophageal junction [GEJ])
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Merkel Cell; Mesothelioma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Stomach Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1, Dose Escalation: INCAGN01949 + Nivolumab (Experimental): INCAGN01949 (70, 200, 350, or 700 milligrams [mg]) combined with nivolumab 240 mg in participants with advanced or metastatic select solid tumors
  Interventions: Drug: INCAGN01949; Drug: Nivolumab
- Phase 1, Dose Escalation: INCAGN01949 + Ipilimumab (Experimental): INCAGN01949 (70, 200, 350, or 700 mg) combined with ipilimumab 1 mg/kilogram (kg) in participants with advanced or metastatic select solid tumors
  Interventions: Drug: INCAGN01949; Drug: Ipilimumab
- Phase 1, Dose Escalation: INCAGN01949 + Nivolumab + Ipilimumab (Experimental): INCAGN01949 combined with nivolumab 3 mg/kg and ipilimumab 1 mg/kg in participants with advanced or metastatic select solid tumors
  Interventions: Drug: INCAGN01949; Drug: Nivolumab; Drug: Ipilimumab
- Phase 1, Safety Expansion: INCAGN01949 + Nivolumab (Experimental): Run-in with INCAGN01949 (70, 200, or 350 mg) x 2 doses, followed by INCAGN01949 (70, 200, or 350 mg) combined with nivolumab 240 mg in participants with advanced or metastatic select solid tumors
  Interventions: Drug: INCAGN01949; Drug: Nivolumab
- Phase 1, Safety Expansion: INCAGN01949 + Nivolumab + Ipilimumab (Experimental): Run-in with INCAGN01949 x 2 doses, followed by INCAGN01949 combined with nivolumab 3 mg/kg and ipilimumab 1 mg/kg in participants with advanced or metastatic select solid tumors
  Interventions: Drug: INCAGN01949; Drug: Nivolumab; Drug: Ipilimumab
- Phase 2, Part A: INCAGN01949 + nivolumab (Experimental): INCAGN01949 combined with nivolumab in programmed cell death protein 1 (PD-1)/programmed cell death protein ligand 1 (PD-L1) refractory participants with gastric cancer, squamous cell carcinoma of the head and neck (SCCHN), non-small cell lung cancer (NSCLC), or renal cell carcinoma (RCC)
  Interventions: Drug: INCAGN01949; Drug: Nivolumab
- Phase 2, Part B: INCAGN01949; INCAGN01949 + nivolumab; INCAGN01949 + nivolumab + ipilimumab (Experimental): INCAGN01949 alone, combined with nivolumab, and combined with nivolumab and ipilimumab in PD-1/L1 refractory participants with advanced or metastatic gastric cancer, SCCHN, NSCLC, or RCC
  Interventions: Drug: INCAGN01949; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: INCAGN01949 — In Phase 1, participants will receive INCAGN01949 administered intravenously (IV) at the protocol-defined dose according to cohort enrollment. In Phase 2, participants will receive INCAGN01949 administered IV at the recommended dose from Phase 1.
Drug: Nivolumab — Nivolumab will be administered IV at the protocol-defined dose according to assigned treatment group.
  Arms: Phase 1, Dose Escalation: INCAGN01949 + Nivolumab; Phase 1, Dose Escalation: INCAGN01949 + Nivolumab + Ipilimumab; Phase 1, Safety Expansion: INCAGN01949 + Nivolumab; Phase 1, Safety Expansion: INCAGN01949 + Nivolumab + Ipilimumab; Phase 2, Part A: INCAGN01949 + nivolumab; Phase 2, Part B: INCAGN01949; INCAGN01949 + nivolumab; INCAGN01949 + nivolumab + ipilimumab
Drug: Ipilimumab — Ipilimumab will be administered IV at the protocol-defined dose according to assigned treatment group.
  Arms: Phase 1, Dose Escalation: INCAGN01949 + Ipilimumab; Phase 1, Dose Escalation: INCAGN01949 + Nivolumab + Ipilimumab; Phase 1, Safety Expansion: INCAGN01949 + Nivolumab + Ipilimumab; Phase 2, Part B: INCAGN01949; INCAGN01949 + nivolumab; INCAGN01949 + nivolumab + ipilimumab

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of INCAGN01949 when given in combination with immune therapies in participants with advanced or metastatic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Phase 1: Subjects with advanced or metastatic solid tumors.
* Phase 1: Subjects who have disease progression after treatment with available therapies.
* Phase 2: Subjects with advanced or metastatic gastric cancer, SCCHN, NSCLC, or RCC and are considered refractory to prior PD-1/L1 therapy.
* Presence of measurable disease based on RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.

Exclusion Criteria:

* Laboratory and medical history parameters not within the Protocol-defined range
* Receipt of anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy.
* Active autoimmune disease.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.
* Known history of human immunodeficiency virus (HIV); HIV 1/2 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Janik, MD, Study Director — Incyte Corporation
Locations (15):
- United States (15):
  - The University of Alabama Birmingham (UAB), Birmingham, Alabama
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Mount Sinai Medical Center of Florida, Inc., Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center At Hackensack UMC, Hackensack, New Jersey
  - Rutgers, The State University, New Brunswick, New Jersey
  - New York University Clinical Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, LLC (SCRI), Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 study centers in the United States in two parts: dose escalation (Part 1) and safety expansion (Part 2).
Groups:
- Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg: Participants with advanced or metastatic select solid tumors received INCAGN01949 70 milligrams (mg) every 2 weeks (Q2W) beginning on Cycle 1 Day 1, followed by nivolumab 240 mg Q2W beginning on Cycle 1 Day 1, administered as intravenous (IV) infusions.
- Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg: Participants with advanced or metastatic select solid tumors received INCAGN01949 200 mg Q2W beginning on Cycle 1 Day 1, followed by nivolumab 240 mg Q2W beginning on Cycle 1 Day 1, administered as IV infusions.
- Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg: Participants with advanced or metastatic select solid tumors received INCAGN01949 350 mg Q2W beginning on Cycle 1 Day 1, followed by nivolumab 240 mg Q2W beginning on Cycle 1 Day 1, administered as IV infusions.
- Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg: Participants with advanced or metastatic select solid tumors received INCAGN01949 700 mg Q2W beginning on Cycle 1 Day 1, followed by nivolumab 240 mg Q2W beginning on Cycle 1 Day 1, administered as IV infusions.
- Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg: Participants with advanced or metastatic select solid tumors received INCAGN01949 70 mg Q2W beginning on Cycle 1 Day 1, followed by ipilimumab 1 mg/kilogram (kg) every 6 weeks (Q6W) beginning on Cycle 1 Day 1, administered as IV infusions.
- Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg: Participants with advanced or metastatic select solid tumors received INCAGN01949 200 mg Q2W beginning on Cycle 1 Day 1, followed by ipilimumab 1 mg/kg Q6W beginning on Cycle 1 Day 1, administered as IV infusions.
- Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg: Participants with advanced or metastatic select solid tumors received INCAGN01949 350 mg Q2W beginning on Cycle 1 Day 1, followed by ipilimumab 1 mg/kg Q6W beginning on Cycle 1 Day 1, administered as IV infusions.
- Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg: Participants with advanced or metastatic select solid tumors received INCAGN01949 700 mg Q2W beginning on Cycle 1 Day 1, followed by ipilimumab 1 mg/kg Q6W beginning on Cycle 1 Day 1, administered as IV infusions.
- Phase 1, Dose Escalation: INCAGN01949 + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg: Participants with advanced or metastatic select solid tumors were to have received INCAGN01949 at the assigned dose level Q2W in combination with nivolumab 3 mg/kg Q2W and ipilimumab 1 mg/kg Q6W, all administered as IV infusions beginning on Cycle 1 Day 1.
- Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg: Participants with advanced or metastatic select solid tumors received INCAGN01949 70 mg Q2W beginning on Cycle 1 Day 1, followed by nivolumab 240 mg Q2W beginning on Cycle 3 Day 1, administered as IV infusions.
- Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg: Participants with advanced or metastatic select solid tumors received INCAGN01949 200 mg Q2W beginning on Cycle 1 Day 1, followed by nivolumab 240 mg Q2W beginning on Cycle 3 Day 1, administered as IV infusions.
- Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg: Participants with advanced or metastatic select solid tumors received INCAGN01949 350 mg Q2W beginning on Cycle 1 Day 1, followed by nivolumab 240 mg Q2W beginning on Cycle 3 Day 1, administered as IV infusions.
- Phase 1, Safety Expansion: INCAGN01949 + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg: Participants with advanced or metastatic solid tumors were to have received INCAGN01949 at the assigned dose level Q2W beginning on Cycle 1 Day 1, in combination with nivolumab 3 mg/kg Q2W beginning on Cycle 3 Day 1 and ipilimumab 1 mg/kg Q6W beginning on Cycle 3 Day 1, administered as IV infusions.
- Phase 2, Part A: INCAGN01949 + Nivolumab: Programmed cell death protein 1 (PD-1)/programmed cell death protein ligand 1 (PD-L1) refractory participants with gastric cancer, squamous cell carcinoma of the head and neck (SCCHN), non-small cell lung cancer (NSCLC), or renal cell carcinoma (RCC) were to have received a range of doses of INCAGN01949 found to be safe in Phase 1 in combination with nivolumab, administered as IV infusions.
- Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab: PD-1/L1 refractory participants with advanced or metastatic gastric cancer, SCCHN, NSCLC, or RCC were to have received a range of doses of INCAGN01949 found to be safe in Phase 1. INCAGN01949 was to have been administered alone, in combination with nivolumab, and in combination with nivolumab and ipilimumab, administered as IV infusions.
Period: Overall Study
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 + Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Started | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 0 (This treatment group did not open for enrollment.) | 6 | 6 | 6 | 0 (This treatment group did not open for enrollment.) | 0 (Phase 2 of the study did not open for enrollment.) | 0 (Phase 2 of the study did not open for enrollment.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 0 | 6 | 6 | 6 | 0 | 0 | 0
Not completed — Death | 3 | 2 | 4 | 4 | 2 | 2 | 3 | 1 | 0 | 5 | 4 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Survival Follow-up No Longer Required per Protocol Amendment | 1 | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg | Total
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 6 | 6 | 6 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (7.53) | 58.0 (3.16) | 60.0 (5.00) | 67.8 (8.07) | 58.5 (6.45) | 60.6 (10.21) | 59.3 (12.71) | 50.0 (20.52) | 60.5 (8.73) | 55.7 (15.96) | 64.0 (13.96) | 58.77 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 2 | 1 | 2 | 3 | 1 | 6 | 3 | 2 | 26
  Male | 1 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 0 | 3 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 4 | 4 | 4 | 3 | 4 | 4 | 3 | 6 | 6 | 6 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 6
  White | 4 | 4 | 4 | 5 | 3 | 3 | 2 | 3 | 5 | 6 | 5 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results that occurred after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any adverse event either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 17.4 months
Population: Full Analysis Set (FAS): all participants enrolled in the study who received ≥ 1 dose of INCAGN01949, nivolumab, or ipilimumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 6 | 6 | 6
Participants | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 6 | 6 | 6

2. Primary Outcome: Phase 1: Number of Participants With a Grade 3 or Higher TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. A TEAE was defined as any adverse event either reported for the first time or the worsening of a pre-existing event after the first dose of study drug. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) v4.03. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death due to AE.
Time Frame: up to 17.4 months
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 6 | 6 | 6
Participants | 2 | 1 | 3 | 3 | 2 | 2 | 3 | 1 | 5 | 4 | 3

3. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1), as determined by investigator assessment of radiographic disease assessments, recorded before and including the first event of progressive disease (PD). CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 24 months
Population: Phase 2 of the study did not open for enrollment.
Arm/Group | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 1: ORR
Description: ORR was defined as the percentage of participants with a confirmed best overall response of CR or PR, per RECIST v1.1, as determined by investigator assessment of radiographic disease assessments, recorded before and including the first event of PD. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 15.6 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 6 | 6 | 6
percentage of participants | 25.0 | 25.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0

5. Secondary Outcome: Phase 1: Duration of Response (DOR)
Description: DOR was defined as the time from the first overall response contributing to a confirmed objective response (CR or PR) to the earlier of the participant's death from any cause or first assessment of PD, determined by investigator assessment of radiographic disease assessments per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 11.0 months
Population: FAS. The confidence interval was calculated using the method of Brookmeyer and Crowley. Only participants with a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg
Number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
days | 97.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |  |  |  |  |  |  |  | 86.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. |

6. Secondary Outcome: Phase 2: DOR
Description: as for outcome 5
Time Frame: up to 24 months
Population: Phase 2 of the study did not open for enrollment.
Arm/Group | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 1: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a CR, PR, or stable disease (SD), determined by investigator assessment of radiographic disease assessments per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 15.6 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 4 | 5 | 4 | 3 | 6 | 6 | 6
percentage of participants | 25.0 | 25.0 | 40.0 | 0.0 | 75.0 | 0.0 | 50.0 | 33.3 | 33.3 | 33.3 | 66.7

8. Secondary Outcome: Phase 2: DCR
Description: DCR was defined as the percentage of participants with a CR, PR, or SD, determined by investigator assessment of radiographic disease assessments per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 24 months
Population: Phase 2 of the study did not open for enrollment.
Arm/Group | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase 1: Duration of Disease Control
Description: Duration of disease control (CR, PR, and SD) was measured from the first report of SD or better until PD or death from any cause, if occurring sooner than progression, determined by investigator assessment of radiographic disease assessments per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. SD: no change in target lesions to qualify for CR, PR, or PD. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 15.4 months
Population: FAS. The confidence interval was calculated based on the exact method for binomial distributions. Only participants with a confirmed CR, PR, or SD were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg
Number analyzed (Participants) | 1 | 1 | 2 | 0 | 3 | 0 | 2 | 1 | 2 | 2 | 4
days | 97.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 120.0 [61.0 to 179.0] |  | 58.0 [43.0 to 113.0] |  | 298.5 [169.0 to 428.0] | 100.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 252.0 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 117.0 [86.0 to 148.0] | 115.0 [52.0 to 418.0]

10. Secondary Outcome: Phase 2: Duration of Disease Control
Description: as for outcome 9
Time Frame: up to 24 months
Population: Phase 2 of the study did not open for enrollment.
Arm/Group | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Phase 1: Progression-free Survival (PFS)
Description: PFS was defined as the length of time between the Baseline visit (Day 1) and the earlier of death or the first assessment of PD, as determined by investigator assessment of objective radiographic disease assessments per RECIST v1.1.
Time Frame: up to 15.6 months
Population: FAS. Median survival time was estimated using the Kaplan-Meier method. The confidence interval was calculated using the method of Brookmeyer and Crowley. Only participants with events of disease progression or death were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4 | 5 | 4 | 3 | 4 | 6 | 6
days | 1.8 [1.0 to 4.9] | 1.8 [1.4 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 2.7 [1.4 to 7.5] | 1.8 [0.8 to 2.1] | 3.5 [0.7 to 5.4] | 1.6 [1.2 to 1.8] | 4.6 [1.2 to 15.7] | 1.8 [1.7 to 5.1] | 1.6 [0.1 to 9.9] | 2.2 [1.8 to 6.7] | 4.6 [1.8 to 15.5]

12. Secondary Outcome: Phase 2: PFS
Description: as for outcome 11
Time Frame: up to 24 months
Population: Phase 2 of the study did not open for enrollment.
Arm/Group | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Phase 2: Number of Participants With TEAEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results that occurred after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any adverse event either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 24 months
Population: Phase 2 of the study did not open for enrollment.
Arm/Group | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Phase 2: Number of Participants With a Grade 3 or Higher TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. A TEAE was defined as any adverse event either reported for the first time or the worsening of a pre-existing event after the first dose of study drug. The severity of AEs was assessed using CTCAE v4.03. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death due to AE.
Time Frame: up to 24 months
Population: Phase 2 of the study did not open for enrollment.
Arm/Group | Phase 2, Part A: INCAGN01949 + Nivolumab | Phase 2, Part B: INCAGN01949; INCAGN01949 + Nivolumab; INCAGN01949 + Nivolumab + Ipilimumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 17.4 months
Description: Treatment-emergent adverse events, defined as any adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug, have been reported.
Groups:
- Total: Total
Arm/Group | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg | Total
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/4 | 4/5 | 4/5 | 2/4 | 2/5 | 3/4 | 1/3 | 5/6 | 4/6 | 3/6 | 33/52
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/4 | 4/5 | 3/5 | 2/4 | 2/5 | 2/4 | 1/3 | 4/6 | 3/6 | 3/6 | 28/52
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 5/5 | 4/4 | 5/5 | 4/4 | 3/3 | 6/6 | 6/6 | 6/6 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg (N=4) | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg (N=4) | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg (N=5) | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg (N=5) | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg (N=4) | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg (N=5) | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg (N=4) | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg (N=3) | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg (N=6) | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg (N=6) | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg (N=6) | Total (N=52)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 11 (11)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 4 (6)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Escalation: INCAGN01949 70 mg + Nivolumab 240 mg (N=4) | Phase 1, Dose Escalation: INCAGN01949 200 mg + Nivolumab 240 mg (N=4) | Phase 1, Dose Escalation: INCAGN01949 350 mg + Nivolumab 240 mg (N=5) | Phase 1, Dose Escalation: INCAGN01949 700 mg + Nivolumab 240 mg (N=5) | Phase 1, Dose Escalation: INCAGN01949 70 mg + Ipilimumab 1 mg/kg (N=4) | Phase 1, Dose Escalation: INCAGN01949 200 mg + Ipilimumab 1 mg/kg (N=5) | Phase 1, Dose Escalation: INCAGN01949 350 mg + Ipilimumab 1 mg/kg (N=4) | Phase 1, Dose Escalation: INCAGN01949 700 mg + Ipilimumab 1 mg/kg (N=3) | Phase 1, Safety Expansion: INCAGN01949 70 mg + Nivolumab 240 mg (N=6) | Phase 1, Safety Expansion: INCAGN01949 200 mg + Nivolumab 240 mg (N=6) | Phase 1, Safety Expansion: INCAGN01949 350 mg + Nivolumab 240 mg (N=6) | Total (N=52)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 10 (12)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 5 (6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 10 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 2 (2) | 9 (11)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (5)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 6 (7)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (7)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 9 (11)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 10 (12)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 6 (7)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 6 (8)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 4 (4) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (5) | 3 (4) | 3 (3) | 27 (30)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Halo vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 7 (11)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersplenism (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (1) | 7 (9)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Mucous membrane disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 3 (3) | 3 (4) | 3 (7) | 19 (26)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular icterus (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (3) | 9 (11)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 5 (7)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 6 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (4) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 14 (17)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea capitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (5) | 10 (13)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Because there was limited clinical efficacy, with 3 confirmed responders, Phase 2 of the study did not open for enrollment. There were no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT03241173/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03241173/SAP_002.pdf